CLINICAL TRIAL: NCT06314932
Title: Role of ultraPROcessed Foods in Modulating the Effect of mEditerraNeAn Diet on Human and Planet hEalth - the PROMENADE Study
Brief Title: Role of Ultra-processed Foods in Modulating the Effect of Mediterranean Diet
Acronym: PROMENADE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: University of Florence (Other); University of Teramo (Other)
Responsible Party: Principal Investigator, Daniela Martini, Associate Professor, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: spe123.23
Record Dates: First submitted 2024-03-01; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Overweight
Keywords: Mediterranean diet; Food processing; Human health; Sustainability
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High UPF (Experimental): Group starting with the Mediterranean diet (MD) high in ultra-processed foods (UPF)
  Interventions: Other: MD high in UPF; Other: MD low in UPF
- Low UPF (Active Comparator): Group starting with the Mediterranean diet (MD) low in ultra-processed foods (UPF)
  Interventions: Other: MD high in UPF; Other: MD low in UPF

INTERVENTIONS:
Other: MD high in UPF — A 3-month dietary intervention with a Mediterranean diet with 5 servings/day of UPF, as defined by the NOVA system (e.g., flavored yogurt, breakfast cereals with added sugar, processed meat).
Other: MD low in UPF — A 3-month dietary intervention with a Mediterranean diet with 5 servings/day of products from the same food group, but non-UPF (e.g., plain yogurt, breakfast cereals with no added sugar, unprocessed meat)

SUMMARY:
Mediterranean diet is worldwide promoted as one of the healthiest and most sustainable dietary patterns. One of the main pillars of Mediterranean diet is the abundant consumption of plant-based ingredients typically consumed as raw or minimally processed. However, even in the Mediterranean countries, these fresh foods are increasingly replaced by ultra-processed foods (UPF). Epidemiological evidence suggests that consumption of UPF may be detrimental to human health, but there is only one clinical trial on this topic which is largely debated in the scientific community due to limitations related to the short duration of the trial and the composition of dietary interventions.

The present study aims at exploring whether the inclusion of UPF within a Mediterranean-based dietary pattern can impact on cardiometabolic markers, gut microbiota and other health markers in a dietary intervention performed in Italian subjects. For this purpose, 50 clinically healthy subjects will be recruited for a 7-month randomized, open, cross-over dietary trial. Eligible participants will be randomly assigned to consume a 3-month Mediterranean diet high in UPF (intervention group) or a low-UPF Mediterranean diet (control group), spaced by a 1-month wash-out period. The two diets will have the same composition in terms of food groups. However, in the high-UPF Mediterranean diet group, 5 servings/day of UPF, as defined by the NOVA system, will be consumed (e.g., flavored yogurt, breakfast cereals with added sugar, processed meat). In the control group, these foods will be replaced by products from the same food group, but not UPF (e.g., plain yogurt, breakfast cereals with no added sugar, unprocessed meat). The inflammatory potential of pairs of food products, both UPF and non UPF, will be evaluated using an in vitro cell model testing the modulation of inflammatory markers. Before and after each intervention blood, urine and fecal samples will be collected. The primary endpoint is change in low-density lipoprotein (LDL) cholesterol levels from baseline. Among the other markers, blood pressure and anthropometric parameters will be measured; biochemical parameters, adipokines, inflammatory and oxidative stress markers, fecal microbiota composition and short chain fatty acids (SCFAs) will be analyzed. Adherence to the study, dietary intake and food waste production will be evaluated through specific food diaries, useful also for estimating the metabolic food waste.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* BMI between 25.0 and 29.9 kg/m2 and the simultaneous presence of at least one of the following criteria, defined by the Guidelines for cardiovascular disease prevention of the European Society of Cardiology:
* total cholesterol levels >190 mg/dL
* LDL-cholesterol levels >115 mg/dL
* triglyceride levels >150 mg/dL
* glucose levels in the range 111-125 mg/dL

Exclusion Criteria:

* presence of current serious illness or unstable condition that requires physician supervision of diet (e.g., recent myocardial infarction, chronic liver disease, inflammatory bowel diseases, renal or digestive disorders)
* pregnancy or intention to become pregnant in the next 12 months
* lactation
* current or recent (past 3 months) use of supplements or antibiotic therapy
* current or recent (past 6 months) adoption of specific restrictive diets (e.g., low-calorie or vegetarian diets)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Low-density lipoprotein (LDL) cholesterol levels | 7 months
  Measurement of LDL-cholesterol levels change from the beginning to the end of each of the two intervention phases in mg/dL

SECONDARY OUTCOMES:
Total cholesterol levels | 7 months
  Measurement of total cholesterol levels change from the beginning to the end of each of the two intervention phases in mg/dL
High-density lipoprotein (HDL) cholesterol levels | 7 months
  Measurement of HDL cholesterol levels change from the beginning to the end of each of the two intervention phases in mg/dL
Triglycerides levels | 7 months
  Measurement of triglyceride levels change from the beginning to the end of each of the two intervention phases in mg/dL
Fasting blood glucose levels | 7 months
  Measurement of fasting blood glucose levels change from the beginning to the end of each of the two intervention phases in mg/dL
Insulin levels | 7 months
  Measurement of insulin levels change from the beginning to the end of each of the two intervention phases in U/I
Aspartate aminotransferase (AST) levels | 7 months
  Measurement of AST levels change from the beginning to the end of each of the two intervention phases in U/I
Alanine aminotransferase (ALT) levels | 7 months
  Measurement of ALT levels change from the beginning to the end of each of the two intervention phases in U/I
Gamma-glutamyl transferase (GGT) levels | 7 months
  Measurement of GGT levels change from the beginning to the end of each of the two intervention phases in U/I
Folates levels | 7 months
  Measurement of folate levels change from the beginning to the end of each of the two intervention phases in ng/mL
Vitamin B12 levels | 7 months
  Measurement of vitamin B12 levels change from the beginning to the end of each of the two intervention phases in pg/mL
Urea levels | 7 months
  Measurement of urea levels change from the beginning to the end of each of the two intervention phases in mg/dL
Creatinine levels | 7 months
  Measurement of creatinine levels change from the beginning to the end of each of the two intervention phases in mg/dL
Body weight | 7 months
  Measurement of body weight change from the beginning to the end of each of the two intervention phases in kg
Body mass index (BMI) | 7 months
  Measurement of BMI change from the beginning to the end of each of the two intervention phases. Weight and height will be combined to report BMI in kg/m^2
Fat mass | 7 months
  Measurement of fat mass change from the beginning to the end of each of the two intervention phases. Percentage of fat mass will be assessed using the Akern bioelectrical impedance analyser (model SE 101).
Concentration of ghrelin in plasma | 7 months
  Measurement of ghrelin change from the beginning to the end of each of the two intervention phases in pg/mL
Concentration of leptin in plasma | 7 months
  Measurement of leptin change from the beginning to the end of each of the two intervention phases in ng/mL
Concentration of adiponectin in plasma | 7 months
  Measurement of adiponectin change from the beginning to the end of each of the two intervention phases in microg/mL
Concentration of resistin in plasma | 7 months
  Measurement of resistin change from the beginning to the end of each of the two intervention phases in ng/mL
Concentration of visfatin in plasma | 7 months
  Measurement of visfatin change from the beginning to the end of each of the two intervention phases in ng/mL
Concentration of interleukin (IL)-4 in plasma | 7 months
  Measurement of IL-4 change from the beginning to the end of each of the two intervention phases in pg/mL
Concentration of interleukin (IL)-6 in plasma | 7 months
  Measurement of IL-6 change from the beginning to the end of each of the two intervention phases in pg/mL
Concentration of interleukin (IL)-10 in plasma | 7 months
  Measurement of IL-10 change from the beginning to the end of each of the two intervention phases in pg/mL
Concentration of Protein C-reactive (PCR) in plasma | 7 months
  Measurement of protein C-reactive (PCR) change from the beginning to the end of each of the two intervention phases in mg/L
Concentration of interferon gamma (IFN-γ) in plasma | 7 months
  Measurement of IFN-γ change from the beginning to the end of each of the two intervention phases in pg/mL
Concentration of tumor necrosis factor -alpha (TNF-α) in plasma | 7 months
  Measurement of TNF-α change from the beginning to the end of each of the two intervention phases in pg/mL
DNA damage expressed as number of DNA strand breaks induced by hydrogen peroxide (H2O2) | 7 months
  Measurement of H2O2-induced DNA strand breaks change from the beginning to the end of each of the two intervention phases in percentage (%)
Concentration of F2-isoprostanes in urine | 7 months
  Measurement of F2-isoprostanes change from the beginning to the end of each of the two intervention phases in pg/mosm
Gut microbiota composition and function changes | 7 months
  Measurement of gut microbiota composition change from the beginning to the end of each of the two intervention phases. Each subject will be asked for a stool sample at the beginning and at the end of each intervention phases in order to analyse the composition of the gut microbiota and short-chain fatty acids production.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Florence, Florence
  - University of Milan, Milan

REFERENCES:
- [Derived] Dinu M, Angelino D, Del Bo' C, Serafini M, Sofi F, Martini D. Role of ultra-processed foods in modulating the effect of Mediterranean diet on human and planet health-study protocol of the PROMENADE randomized controlled trial. Trials. 2024 Sep 30;25(1):641. doi: 10.1186/s13063-024-08470-6. PMID 39350201